CLINICAL TRIAL: NCT06606197
Title: CRIBADO DE VIRUS DE LA HEPATITIS C en Hombres Que Tienen Sexo Con Hombres (HSH) Sitges
Brief Title: Hepatitis C Prevalence in Men Who Have Sex With Men
Status: Completed | Type: Observational
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Other Study IDs: CSAPG_34
Record Dates: First submitted 2024-09-16; First posted 2024-09-20 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-09

CONDITIONS: Hepatitis C
Keywords: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men who have sex with men
  Interventions: Other: Having sex with other men

INTERVENTIONS:
Other: Having sex with other men — Having sex with other men

SUMMARY:
This is an observational study aimed at determining the prevalence of hepatitis C in a specific population: men who have sex with men.

ELIGIBILITY:
Inclusion Criteria:

* Having sex with men

Exclusion Criteria:

* Refusal to participate in the trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men
Study Population: Population attending the "International Bears Sitges Week" festival in September 2022 in Sitges, Barcelona.
Sampling Method: Non-Probability Sample
Enrollment: 454 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2022-09-11 (Actual); Study Completion 2022-09-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with Hepatitis C screening positive | Baseline
  A positive result will be defined as a positive outcome in both the serological test and the viral load test

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Albertos, MD, Principal Investigator — CSAPG
Locations (1):
- Consorci Sanitari Alt Penedès Garraf, Vilafranca del Penedès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol, ICF
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.

REFERENCES:
- [Result] Albertos S, Majo FX, Esteban R, Colom J, Buti M. A large-scale screening of hepatitis C among men who have sex with men in the community using saliva point-of-care testing. Front Public Health. 2024 Dec 9;12:1478195. doi: 10.3389/fpubh.2024.1478195. eCollection 2024. PMID 39717035
- See also: Trial results — https://pubmed.ncbi.nlm.nih.gov/39717035/